CLINICAL TRIAL: NCT00254033
Title: The Role of the Dopaminergic Brain Reward System in Apathy Associated With Alzheimer's Disease
Brief Title: Apathy Associated With Alzheimer's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: American Health Assistance Foundation (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 065-2003; AHAF Grant Number: A2003-236
Record Dates: First submitted 2005-11-10; First posted 2005-11-15 (Estimated); Last update posted 2017-04-28 (Actual); Status verified 2017-04

CONDITIONS: Dementia; Alzheimer Disease
Keywords: Alzheimer's Disease; Apathy; Brain Reward System; Dopamine; Dextroamphetamine Challenge; Methylphenidate
MeSH Terms: conditions — Dementia; Alzheimer Disease; Lethargy | interventions — Dextroamphetamine; Methylphenidate

INTERVENTIONS:
Drug: Dextroamphetamine
Drug: Methylphenidate

SUMMARY:
Apathy, or lack of motivation, affects up to 80% of Alzheimer's disease (AD) patients. These amotivational symptoms increase patient reliance on caregivers, increase caregiver burden and distress, and increase the risk of patient institutionalization. Only 50% of patients with apathy respond to current treatment with cholinesterase inhibitors. The mechanism of apathy in AD is unknown hampering rational treatment. Our proposed pilot study will provide initial data required to develop an amphetamine challenge paradigm to probe the brain reward system. These results will be used to develop a larger study evaluating the role of the brain reward system in apathy in AD and link this information with pharmacologic treatment. AD is a complex neurobiological illness that needs to be understood at several levels to optimize treatment. At a neurochemical level, one has to identify the neurotransmitter abnormalities that accompany the clinical symptoms. The neurochemical level of analysis provides the link between pathology and symptoms and, for now, is the only avenue for biological therapies. Next, one has to translate knowledge of neurochemical abnormalities to practical treatments for the symptoms of AD. This pilot will allow us to develop a study that can address both of these goals. Furthermore, the larger study will further define the emerging concept of apathy as a syndrome and has broader implications for apathy in many other neuropsychiatric diseases.

ELIGIBILITY:
Inclusion Criteria:

* age > 55 years
* meet DSM-IV criteria for primary degenerative dementia
* meet NINCDS-ARDA criteria for probable Alzheimer's Disease of at least one year's duration
* mild to moderate cognitive impairment (Global Deterioration Scale GDS <6, Mini-Mental State Examination >10
* on a stable dose of a cholinesterase inhibitor for at least 3 months
* apathetic group only: Neuropsychiatric Inventory (NPI) Apathy subscale score >=2

Exclusion Criteria:

* abnormal biochemical screening: blood cell count, vitamin B12, thyroid function tests, and syphilis screening tests
* significant medical illness or other medical/neurological conditions which diminish cognitive function
* evidence of seizure disorder
* an Hachinski ischemic score >3 indicating vascular dementia
* a brain computed tomographic (CT) scan revealing focal lesions, or inconsistent with AD
* electrocardiographic, laboratory or physical evidence of significant cardiovascular disease
* presence of premorbid or current psychiatric diagnosis including: major depression, schizophrenia, psychotic symptoms of a severity likely to provoke violent or dangerous behaviour (i.e., command hallucinations to harm people or persecutory delusions that provoke violent reactions)
* current or past psychoactive substance abuse or dependence (including alcohol, excluding nicotine)
* contraindications to receiving dextroamphetamine or methylphenidate
* have had administration of a depot neuroleptic injection within one treatment cycle of the first visit

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2003-10; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
Addiction Research Centre Inventory (ARCI)
Apathy Evaluation Scale-Caregiver (AES-C)

SECONDARY OUTCOMES:
Profile of Mood States (POMS)
Continuous Performance Test (CPT)
Neuropsychiatric Inventory (NPI)

CONTACTS AND LOCATIONS:
Overall Officials: Krista L Lanctot, PhD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Result] Lanctot KL, Herrmann N, Black SE, Ryan M, Rothenburg LS, Liu BA, Busto UE. Apathy associated with Alzheimer disease: use of dextroamphetamine challenge. Am J Geriatr Psychiatry. 2008 Jul;16(7):551-7. doi: 10.1097/JGP.0b013e318170a6d1. PMID 18591575